CLINICAL TRIAL: NCT06147687
Title: FEMaLe: The Use of Machine Learning for Early Diagnosis of Endometriosis Based on Patient Self-reported Data - Study Protocol of a Multicenter Trial
Brief Title: Machine Learning for Early Diagnosis of Endometriosis(MLEndo)
Acronym: MLEndo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Semmelweis University (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Semmelweis
Record Dates: First submitted 2023-09-25; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis; Pelvic Pain; Infertility, Female
Keywords: endometriosis; infertility
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Infertility, Female; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with endometriosis and Healthy controls: 5 000 people with endometriosis will be enrolled and followed up for 1one year. To participate in the study, the women must meet the inclusion criteria.
  Interventions: Diagnostic Test: Self reported data collection
- Control: 5 000 people in a control group will be enrolled and followed up for 1one year. To participate in the study, the women must meet the inclusion criteria.
  Interventions: Diagnostic Test: Self reported data collection

INTERVENTIONS:
Diagnostic Test: Self reported data collection — ML assessement of colleceted data
  Other Names: ML assessement

SUMMARY:
The project aims to create a large prospective data bank using the Lucy medical mobile application and collect and analyze patient profiles and structured clinical data with artificial intelligence. In addition, authors will investigate the association of removed or restricted dietary components with quality of life, pain, and central sensitization.

DETAILED DESCRIPTION:
Introduction: Endometriosis is a complex and chronic disease that affects ∼176 million women of reproductive age and remains largely unresolved. It is defined by the presence of endometrium-like tissue outside the uterus and is commonly associated with chronic pelvic pain, infertility, and decreased quality of life. Despite numerous proposed screening and triage methods such as biomarkers, genomic analysis, imaging techniques, and questionnaires to replace invasive diagnostic laparoscopy, none have been widely adopted in clinical practice.

. Despite the availability of various screening methods (e.g., biomarkers, genomic analysis, imaging techniques) that are intended to replace the need for invasive diagnostic laparoscopy, the time to diagnosis remains in the range of 4 to 11 years. Aims: The project aims to create a large prospective data bank using the Lucy medical mobile application and collect and analyze patient profiles and structured clinical data with artificial intelligence. In addition, authors will investigate the association of removed or restricted dietary components with quality of life, pain, and central sensitization. Methods: A Baseline and Longitudinal Questionnaire in the Lucy app collects self-reported information on symptoms related to endometriosis, socio-demographics, mental and physical health, nutritional, and other lifestyle factors. 5,000 women with endometriosis and 5,000 women in a control group will be enrolled and followed up for one year. With this information, any connections between symptoms and endometriosis will be analyzed with machine learning. Conclusions: Authors can develop a phenotypic description of women with endometriosis by linking the collected data with existing registry-based information on endometriosis diagnosis, healthcare utilization, and big data approach. This may help to achieve earlier detection of endometriosis with pelvic pain and significantly reduce the current diagnostic delay. Additionally, authors can identify nutritional components that may worsen the quality of life and pain in women with endometriosis; thus, authors can create evidence-based dietary recommendations.

Keywords: Endometriosis, Machine learning, Non-invasive diagnosis, Diet

ELIGIBILITY:
Inclusion Criteria:

* Women in reproductive age
* 5000 patients with endometriosis
* 5000 patients without endometriosis

Exclusion Criteria:

* Ongoing pregnancy
* Malignant condition of ovary/uterus/breast

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women suffering from endometriosis and healthy controls
Study Population: 5000/5000 patienets with/without endometriosis This study is conducted as a multicenter, parallel-group trial. Study participants are being recruited through the Lucy app. Data are collected in the following countries: Hungary, Denmark, Sweden, Germany, and Austria. Participant recruitment began in December 2021 and is expected to continue until December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient- profiling using the Lucy app | 24 month
  Establish a comprehensive and extensive prospective big data repository using the Lucy app. This initiative aims to identify unique clinical cohorts by leveraging various factors such as digital footprints, symptoms, patient experiences, comorbidities, clinical severity, and lifestyle patterns. By employing Using ML for big data analysis, authors can build patient profiles and structured clinical data that facilitate the early detection of endometriosis with pelvic pain.
  Self-reported data of the participants will be measured as follows:
  * Evaluating the quality of life using the 5-level EQ-5D (EQ-5D-5L)
  * Endometriosis Health Profile 5 (EHP-5) .
  * Pain scores using the Visual Analogue Scale (VAS) .
  * Central pain sensitization using the short version of Central Sensitization Inventory (CSI-9)

SECONDARY OUTCOMES:
Impact of diet and lifestyle on the development of endometriosis | 24 month
  Additionally, authors can identify nutritional components that may worsen the quality of life and pain in women with endometriosis; thus, they can create evidence-based dietary recommendations.
  The changes in quality of life will be assessed by using Self-reported data of the participants will be measured as follows:
  Change From Baseline in Pain Scores on the Visual Analog Scale at 12 months. Changes from baseline values on EHP5 at 12 months

OTHER OUTCOMES:
Economical burden of endometriosis | 24 month
  Economical burden taking into account the cost of diet and healthcare use. The exact cost of endometriosis related diet will be reported per month in EUR.

CONTACTS AND LOCATIONS:
Overall Officials: Attila Bokor, Principal Investigator — Semmelweis University
Locations (2):
- Hungary (2):
  - Bokor Attila, Budapest
  - Semmelweis University, Budapest

IPD SHARING:
Plan to Share IPD: Yes
In case of any interest we are happy to share IPD
Supporting Information: Study Protocol
Time Frame: Data will become available from 01.01.2025 for 5 years
Access Criteria: Data will be available for researchers in the field